CLINICAL TRIAL: NCT03276754
Title: IMMUNIZATION TO PREVENT ACUTE COPD EXACERBATIONS (IMPACE STUDY)
Brief Title: Immunization To Prevent Acute COPD Exacerbations
Status: Terminated | Type: Observational
Why Stopped: The study was terminated prematurely due to the inability to recruit the planned number of subjects and the interim analysis indicated that the number of included patients did not allow draw any valid conclusion about the main objective of the study
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1851177; IMPACE (Other: Alias Study Number)
Record Dates: First submitted 2017-09-06; First posted 2017-09-08 (Actual); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Pneumococcal Infections; COPD
Keywords: Pneumococcal infections; COPD exacerbations
MeSH Terms: conditions — Pneumococcal Infections; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Prospective multicenter observational study, to evaluate the impact of routine clinical practice vaccination with PCV13 on the reduction of the risk of moderate/severe COPD exacerbations

DETAILED DESCRIPTION:
Patients with chronic obstructive pulmonary disease (COPD) have been demonstrated to have an increased risk of pneumococcal disease. Pneumonia is frequent among patients hospitalized for COPD exacerbations and is associated with increased health care utilization and higher mortality. Up to 50%-70% of exacerbations can be attributed to respiratory infections by viruses or bacteria, even more in the most severe patients. They are often associated with the colonization of airways by multiple bacteria or viruses of low virulence that in normal conditions are parts of the normal flora of the upper airway. Current recommendations for immunization of patients with COPD include vaccination against influenza and Streptococcus pneumoniae. The aim of this study is to evaluate the potential benefits of immunization of COPD patients with PCV13 and/or against influenza in terms of clinical benefits and quality of life.

ELIGIBILITY:
Inclusion criteria:

1. Patient ≥18 years diagnosed with COPD (any stage, the subgroups for the analysis would be based on COPD severity grade)
2. Ability to understand and complete the required QoL questionnaires
3. At least 2 years of clinical history available that includes records of previous moderate/severe exacerbations, influenza and pneumococcal vaccination history comorbidities and previous treatments.
4. Spirometry data (maximum 6 months old, or if not available at enrollment, to be performed as per normal clinical practice at visit 1 +/- one month)

Exclusion criteria:

1. Impossibility to perform prospective follow up
2. Present any immunocompromising condition
3. Present any other respiratory diseases as co-morbidity (subjects with overlap syndromes COPD-asthma will be excluded. Mixed phenotype defined as: symptoms of increased variability of airflow and incompletely reversible airflow obstruction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects ≥18 years diagnosed with COPD, followed up at the Pulmonology Department of the partipant centres
Sampling Method: Probability Sample
Enrollment: 530 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- Spain (11):
  - Hospital Universitario Son Espases, Palma, Balearic Islands
  - Hospital Universitari Mutua Terrassa, Terrassa, Barcelona
  - Hospital el Bierzo, Ponferrada, LEÓN
  - Hospital Universitario Fundacion Alcorcon, Alcorcón, Madrid
  - Hospital Clinico de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Gregorio Marañon, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Complejo Asistencial de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1851177

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants diagnosed with Chronic Obstructive Pulmonary Disease (COPD) across 11 hospitals in Spain were followed up during their routine follow-up visits in this prospective observational study. Participants were prescribed therapies in line with routine clinical practice.
Pre-assignment Details: A total of 530 evaluable participants were included in the study.
Groups:
- Participants With COPD: Participants with COPD having at least 2 years of prior medical record including history of moderate/severe exacerbations, influenza and pneumococcal vaccination history, comorbidities and previous treatments were observed in this prospective study.
  Participants were prescribed therapies in line with routine clinical practice.
Period: Overall Study
Arm/Group | Participants With COPD
Started | 530
Without Pneumococcal Vaccination | 126
With Pneumococcal Vaccination | 404 (Participants with pneumococcal vaccination may include participants with PCV13 vaccine)
13-Valent Pneumococcal Conjugate Vaccine (PCV13) Population | 114
Completed | 421
Not Completed | 109
Not completed — Withdrawal of informed consent | 4
Not completed — Presence of any immunosuppressive condition | 8
Not completed — Lost to Follow-up | 27
Not completed — No data reported at Month 24 | 31
Not completed — Death | 39

BASELINE CHARACTERISTICS:
Population: Analysis population included all evaluable participants whose data were included and prospectively observed in the study.
Arm/Group | Participants With COPD
Number analyzed (Participants) | 530
Age, Continuous [Mean (Standard Deviation); unit: Years] — Overall number of participants, with pneumococcal vaccination, without pneumococcal vaccination and PCV13 population is presented. Population: Number Analyzed signifies number of participants evaluable for the specified rows.
  Years
    Overall | 70.2 (7.9)
    Without pneumococcal vaccination: number analyzed (Participants) | 126
    Without pneumococcal vaccination | 68.2 (8.4)
    With pneumococcal vaccination: number analyzed (Participants) | 404
    With pneumococcal vaccination | 70.8 (7.7)
    PCV13 Population: number analyzed (Participants) | 114
    PCV13 Population | 69.2 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Overall number of participants, with pneumococcal vaccination, without pneumococcal vaccination and PCV13 population is presented. Population: Number Analyzed signifies number of participants evaluable for the specified rows.
  Participants
    Overall: Female | 133
    Overall: Male | 397
    Without pneumococcal vaccination: number analyzed (Participants) | 126
    Without pneumococcal vaccination: Female | 42
    Without pneumococcal vaccination: Male | 84
    With pneumococcal vaccination: number analyzed (Participants) | 404
    With pneumococcal vaccination: Female | 91
    With pneumococcal vaccination: Male | 313
    PCV13 Population: number analyzed (Participants) | 114
    PCV13 Population: Female | 26
    PCV13 Population: Male | 88
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Mean (Standard Deviation); unit: Kilogram] — Overall number of participants, with pneumococcal vaccination, without pneumococcal vaccination and PCV13 population is presented. Population: Number Analyzed signifies number of participants evaluable for the specified rows.
  Kilogram
    Overall: number analyzed (Participants) | 529
    Overall | 75.0 (16.1)
    Without pneumococcal vaccination: number analyzed (Participants) | 126
    Without pneumococcal vaccination | 74.1 (18.9)
    With pneumococcal vaccination: number analyzed (Participants) | 403
    With pneumococcal vaccination | 75.2 (15.1)
    PCV13 Population: number analyzed (Participants) | 114
    PCV13 Population | 75.2 (14.1)
Height [Mean (Standard Deviation); unit: Centimeters] — Overall number of participants, with pneumococcal vaccination, without pneumococcal vaccination and PCV13 population is presented. Population: Number Analyzed signifies number of participants evaluable for the specified rows.
  Centimeters
    Overall | 164.7 (8.4)
    Without pneumococcal vaccination: number analyzed (Participants) | 126
    Without pneumococcal vaccination | 163.8 (9.2)
    With pneumococcal vaccination: number analyzed (Participants) | 404
    With pneumococcal vaccination | 164.9 (8.1)
    PCV13 Population: number analyzed (Participants) | 114
    PCV13 Population | 164.9 (7.9)
Body Mass Index [Mean (Standard Deviation); unit: Kilograms per meter square] — BMI was calculated automatically based on the reported weight and height in the unit of kilograms over squared meters (kg/m^2). Overall number of participants, with pneumococcal vaccination, without pneumococcal vaccination and PCV13 population is presented. Population: Number Analyzed signifies number of participants evaluable for the specified rows.
  Kilograms per meter square
    Overall: number analyzed (Participants) | 529
    Overall | 27.5 (5.1)
    Without pneumococcal vaccination: number analyzed (Participants) | 126
    Without pneumococcal vaccination | 27.4 (5.8)
    With pneumococcal vaccination: number analyzed (Participants) | 403
    With pneumococcal vaccination | 27.6 (4.8)
    PCV13 Population: number analyzed (Participants) | 114
    PCV13 Population | 27.7 (4.8)
Waist circumference [Mean (Standard Deviation); unit: Centimeters] — Overall number of participants, with pneumococcal vaccination, without pneumococcal vaccination and PCV13 population is presented. Population: Number Analyzed signifies number of participants evaluable for the specified rows.
  Centimeters
    Overall: number analyzed (Participants) | 468
    Overall | 98.4 (16.4)
    Without pneumococcal vaccination: number analyzed (Participants) | 110
    Without pneumococcal vaccination | 99.1 (17.5)
    With pneumococcal vaccination: number analyzed (Participants) | 358
    With pneumococcal vaccination | 98.2 (16.1)
    PCV13 Population: number analyzed (Participants) | 104
    PCV13 Population | 100.1 (17.0)
Relevant Medical History [Count of Participants; unit: Participants] — The participants were reported with the medical history of Yes/No. In case of "Yes" medical history, the following comorbidities were reported: arterial hypertension, dyslipidemia, diabetes mellitus, history of neoplasm, ischemic heart disease, pneumonias in the last year, cardiac failure, chronic renal failure and metabolic syndromes. Overall number of participants, with pneumococcal vaccination, without pneumococcal vaccination and PCV13 population is presented. Population: Number Analyzed signifies number of participants evaluable for the specified rows.
  Participants
    Overall: Medical History- No | 39
    Overall: Medical History- Yes | 491
    Overall: Medical History- Yes (Arterial hypertension) | 279
    Overall: Medical History- Yes (Dyslipidemia) | 241
    Overall: Medical History- Yes (Diabetes mellitus) | 112
    Overall: Medical History- Yes (History of neoplasm) | 78
    Overall: Medical History- Yes (Ischemic heart disease) | 53
    Overall: Medical History- Yes (Cardiac failure) | 37
    Overall: Medical History- Yes (Pneumonias in the last year) | 36
    Overall: Medical History- Yes (Chronic renal failure) | 27
    Overall: Medical History- Yes (Metabolic syndrome) | 2
    Without Pneumococcal Vaccination: No: number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: No | 12
    Without Pneumococcal Vaccination: Yes: number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Yes | 114
    Without Pneumococcal Vaccination: Yes (Arterial hypertension): number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Yes (Arterial hypertension) | 60
    Without Pneumococcal Vaccination: Yes (Dyslipidemia): number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Yes (Dyslipidemia) | 53
    Without Pneumococcal Vaccination: Yes (Diabetes mellitus): number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Yes (Diabetes mellitus) | 27
    Without Pneumococcal Vaccination: Yes (History of neoplasm): number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Yes (History of neoplasm) | 10
    Without Pneumococcal Vaccination: Yes (Ischemic heart disease): number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Yes (Ischemic heart disease) | 6
    Without Pneumococcal Vaccination: Yes (Cardiac failure): number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Yes (Cardiac failure) | 11
    Without Pneumococcal Vaccination: Yes (Pneumonias in the last year): number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Yes (Pneumonias in the last year) | 9
    Without Pneumococcal Vaccination: Yes (Chronic renal failure): number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Yes (Chronic renal failure) | 1
    Without Pneumococcal Vaccination: Yes (Metabolic syndrome): number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Yes (Metabolic syndrome) | 0
    With Pneumococcal Vaccination: No: number analyzed (Participants) | 404
    With Pneumococcal Vaccination: No | 27
    With Pneumococcal Vaccination: Yes: number analyzed (Participants) | 404
    With Pneumococcal Vaccination: Yes | 377
    With Pneumococcal Vaccination: Yes (Arterial hypertension): number analyzed (Participants) | 404
    With Pneumococcal Vaccination: Yes (Arterial hypertension) | 219
    With Pneumococcal Vaccination: Yes (Dyslipidemia): number analyzed (Participants) | 404
    With Pneumococcal Vaccination: Yes (Dyslipidemia) | 188
    With Pneumococcal Vaccination: Yes (Diabetes mellitus): number analyzed (Participants) | 404
    With Pneumococcal Vaccination: Yes (Diabetes mellitus) | 85
    With Pneumococcal Vaccination: Yes (History of neoplasm): number analyzed (Participants) | 404
    With Pneumococcal Vaccination: Yes (History of neoplasm) | 68
    With Pneumococcal Vaccination: Yes (Ischemic heart disease): number analyzed (Participants) | 404
    With Pneumococcal Vaccination: Yes (Ischemic heart disease) | 47
    With Pneumococcal Vaccination: Yes (Cardiac failure): number analyzed (Participants) | 404
    With Pneumococcal Vaccination: Yes (Cardiac failure) | 26
    With Pneumococcal Vaccination: Yes (Pneumonias in the last year): number analyzed (Participants) | 404
    With Pneumococcal Vaccination: Yes (Pneumonias in the last year) | 27
    With Pneumococcal Vaccination: (Chronic renal failure): number analyzed (Participants) | 404
    With Pneumococcal Vaccination: (Chronic renal failure) | 26
    With Pneumococcal Vaccination: (Metabolic syndrome): number analyzed (Participants) | 404
    With Pneumococcal Vaccination: (Metabolic syndrome) | 2
    PCV 13 Population: No: number analyzed (Participants) | 114
    PCV 13 Population: No | 13
    PCV 13 Population: Yes: number analyzed (Participants) | 114
    PCV 13 Population: Yes | 101
    PCV 13 Population: Yes (Arterial hypertension): number analyzed (Participants) | 114
    PCV 13 Population: Yes (Arterial hypertension) | 56
    PCV 13 Population: Yes (Dyslipidemia): number analyzed (Participants) | 114
    PCV 13 Population: Yes (Dyslipidemia) | 53
    PCV 13 Population: Yes (Diabetes mellitus): number analyzed (Participants) | 114
    PCV 13 Population: Yes (Diabetes mellitus) | 23
    PCV 13 Population: Yes (History of neoplasm): number analyzed (Participants) | 114
    PCV 13 Population: Yes (History of neoplasm) | 13
    PCV 13 Population: Yes (Ischemic heart disease): number analyzed (Participants) | 114
    PCV 13 Population: Yes (Ischemic heart disease) | 11
    PCV 13 Population: Yes (Pneumonias in the last year): number analyzed (Participants) | 114
    PCV 13 Population: Yes (Pneumonias in the last year) | 9
    PCV 13 Population: Yes (Cardiac failure): number analyzed (Participants) | 114
    PCV 13 Population: Yes (Cardiac failure) | 2
    PCV 13 Population: Yes (Chronic renal failure): number analyzed (Participants) | 114
    PCV 13 Population: Yes (Chronic renal failure) | 1
Smoking habit [Count of Participants; unit: Participants] — The participants were classified as regular smoker (currently smokes tobacco daily), occasional smoker (does not smoke daily), non-smoker (has not been exposed to smoking) and former smoker (has quit smoking more than 6 months ago). Overall number of participants, with pneumococcal vaccination, without pneumococcal vaccination and PCV13 population is presented. Population: Number Analyzed signifies number of participants evaluable for the specified rows.
  Participants
    Overall: Regular smoker | 98
    Overall: Occasional smoker | 18
    Overall: Non-smoker | 6
    Overall: Former smoker | 408
    Without Pneumococcal Vaccination: number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Regular smoker | 41
    Without Pneumococcal Vaccination: Occasional smoker | 7
    Without Pneumococcal Vaccination: Non-smoker | 0
    Without Pneumococcal Vaccination: Former smoker | 78
    With Pneumococcal Vaccination: number analyzed (Participants) | 404
    With Pneumococcal Vaccination: Regular smoker | 57
    With Pneumococcal Vaccination: Occasional smoker | 11
    With Pneumococcal Vaccination: Non-smoker | 6
    With Pneumococcal Vaccination: Former smoker | 330
    PCV13 Population: number analyzed (Participants) | 114
    PCV13 Population: Regular smoker | 25
    PCV13 Population: Occasional smoker | 3
    PCV13 Population: Non-smoker | 2
    PCV13 Population: Former smoker | 84
Alcohol consumption [Count of Participants; unit: Participants] — The participants were reported with consumption of alcohol as Yes/No. The intake of at least 80 gram/day in the previous year is considered as Yes. Overall number of participants, with pneumococcal vaccination, without pneumococcal vaccination and PCV13 population is presented. Population: Number Analyzed signifies number of participants evaluable for the specified rows.
  Participants
    Overall: No | 511
    Overall: Yes | 19
    Without Pneumococcal Vaccination: number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: No | 118
    Without Pneumococcal Vaccination: Yes | 8
    With Pneumococcal Vaccination: number analyzed (Participants) | 404
    With Pneumococcal Vaccination: No | 393
    With Pneumococcal Vaccination: Yes | 11
    PCV13 Population: number analyzed (Participants) | 114
    PCV13 Population: No | 112
    PCV13 Population: Yes | 2
Forced Expiratory Volume (FEV1) [Mean (Standard Deviation); unit: Percentage] — FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. It is expressed as volume (in milliliters) and is considered normal when it is greater than 80 percent (%) of its theoretical value. Overall number of participants, with pneumococcal vaccination, without pneumococcal vaccination and PCV13 population is presented. Population: Number Analyzed signifies number of participants evaluable for the specified rows.
  Percentage
    Overall: number analyzed (Participants) | 499
    Overall | 53.4 (18.6)
    Without Pneumococcal Vaccination: number analyzed (Participants) | 113
    Without Pneumococcal Vaccination | 52.1 (19.9)
    With Pneumococcal Vaccination: number analyzed (Participants) | 386
    With Pneumococcal Vaccination | 53.8 (18.2)
    PCV13 Population: number analyzed (Participants) | 99
    PCV13 Population | 51.9 (19.0)
Forced Vital Capacity (FVC) [Mean (Standard Deviation); unit: Percentage] — FVC is the volume of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. It is expressed as volume (in ml) and is considered normal when it is greater than 80% of its theoretical value. Overall number of participants, with pneumococcal vaccination, without pneumococcal vaccination and PCV13 population is presented. Population: Number Analyzed signifies number of participants evaluable for the specified rows.
  Percentage
    Overall: number analyzed (Participants) | 499
    Overall | 83.0 (21.4)
    Without Pneumococcal Vaccination: number analyzed (Participants) | 113
    Without Pneumococcal Vaccination | 82.3 (22.4)
    With Pneumococcal Vaccination: number analyzed (Participants) | 386
    With Pneumococcal Vaccination | 83.2 (21.2)
    PCV13 Population: number analyzed (Participants) | 99
    PCV13 Population | 84.5 (22.1)
FEV1/FVC Ratio [Mean (Standard Deviation); unit: Percentage] — FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. FVC is the volume of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. Overall number of participants, with pneumococcal vaccination, without pneumococcal vaccination and PCV13 population is presented. Population: Number Analyzed signifies number of participants evaluable for the specified rows.
  Percentage
    Overall: number analyzed (Participants) | 499
    Overall | 49.3 (11.3)
    Without Pneumococcal Vaccination: number analyzed (Participants) | 113
    Without Pneumococcal Vaccination | 49.5 (12.1)
    With Pneumococcal Vaccination: number analyzed (Participants) | 386
    With Pneumococcal Vaccination | 49.2 (11.0)
    PCV13 Population: number analyzed (Participants) | 99
    PCV13 Population | 48.0 (12.8)
COPD severity (GOLD) [Count of Participants; unit: Participants] — COPD severity in terms Global Initiative for Chronic Obstructive Lung Disease (GOLD) is defined as follows: Grade 1: Mild/unknown (FEV1 greater than equal to [>=]80%, FEV1/FVC Less than [< 0.7] or no spirometry data); Grade 2: Moderate (50% less than equal to [<=] FEV1< 80%,FEV1/FVC < 0.7); Grade 3: Severe (30% <= FEV1 < 50%, FEV1/FVC < 0.7) and Grade 4: Very severe (FEV1< 30% FEV1< 50% plus respiratory failure,FEV1/FVC < 0.7). Overall number of participants, with pneumococcal vaccination, without pneumococcal vaccination and PCV13 population is presented. Population: Number Analyzed signifies number of participants evaluable for the specified rows.
  Participants
    Overall: Grade 1: Mild/unknown | 55
    Overall: Grade 2: Moderate | 218
    Overall: Grade 3: Severe | 178
    Overall: Grade 4: Very severe | 79
    Without Pneumococcal Vaccination: number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Grade 1: Mild/unknown | 14
    Without Pneumococcal Vaccination: Grade 2: Moderate | 44
    Without Pneumococcal Vaccination: Grade 3: Severe | 50
    Without Pneumococcal Vaccination: Grade 4: Very severe | 18
    With Pneumococcal Vaccination: number analyzed (Participants) | 404
    With Pneumococcal Vaccination: Grade 1: Mild/unknown | 41
    With Pneumococcal Vaccination: Grade 2: Moderate | 174
    With Pneumococcal Vaccination: Grade 3: Severe | 128
    With Pneumococcal Vaccination: Grade 4: Very severe | 61
    PCV13 Population: number analyzed (Participants) | 114
    PCV13 Population: Grade 1: Mild/unknown | 12
    PCV13 Population: Grade 2: Moderate | 47
    PCV13 Population: Grade 3: Severe | 36
    PCV13 Population: Grade 4: Very severe | 19
Number of moderate/severe exacerbations prior to study inclusion [Mean (Standard Deviation); unit: Exacerbation per participant in 24 month] — Overall number of participants, with pneumococcal vaccination, without pneumococcal vaccination and PCV13 population is presented. Population: Number Analyzed signifies number of participants evaluable for the specified rows.
  Exacerbation per participant in 24 month
    Overall | 3.3 (3.2)
    Without Pneumococcal Vaccination: number analyzed (Participants) | 126
    Without Pneumococcal Vaccination | 2.9 (2.7)
    With Pneumococcal Vaccination: number analyzed (Participants) | 404
    With Pneumococcal Vaccination | 3.5 (3.3)
    PCV13 Population: number analyzed (Participants) | 114
    PCV13 Population | 2.4 (1.6)
Pneumococcal vaccination prior to study inclusion [Count of Participants; unit: Participants] — The Participants were classified as No (Without pneumococcal vaccination) and Yes (With pneumococcal vaccination). If Yes, then according to the type of pneumococcal vaccination received as: Polysaccharide only (PPSV23 [23 valent pneumococcal polysaccharide vaccine
  ]), Polysaccharide (PPSV23) + Conjugate (PCV13) and Conjugate only (PCV13). Overall number of participants, with pneumococcal vaccination and without pneumococcal vaccination is presented. Population: Number Analyzed signifies number of participants evaluable for the specified rows.
  Participants
    Overall: No | 126
    Overall: Yes | 404
    Overall: Yes, Polysaccharide only (PPSV23) | 180
    Overall: Yes, Polysaccharide (PPSV23) + Conjugate (PCV13) | 142
    Overall: Yes, Conjugate only (PCV13) | 82
    Without pneumococcal vaccination: No: number analyzed (Participants) | 126
    Without pneumococcal vaccination: No | 126
    Without pneumococcal vaccination: Yes: number analyzed (Participants) | 126
    Without pneumococcal vaccination: Yes | 0
    Without pneumococcal vaccination: Yes, Polysaccharide only (PPSV23): number analyzed (Participants) | 126
    Without pneumococcal vaccination: Yes, Polysaccharide only (PPSV23) | 0
    Without pneumococcal vaccination: Yes, Polysaccharide (PPSV23) + Conjugate (PCV13): number analyzed (Participants) | 126
    Without pneumococcal vaccination: Yes, Polysaccharide (PPSV23) + Conjugate (PCV13) | 0
    Without pneumococcal vaccination: Yes, Conjugate only (PCV13): number analyzed (Participants) | 126
    Without pneumococcal vaccination: Yes, Conjugate only (PCV13) | 0
    With pneumococcal vaccination: No: number analyzed (Participants) | 404
    With pneumococcal vaccination: No | 0
    With pneumococcal vaccination: Yes: number analyzed (Participants) | 404
    With pneumococcal vaccination: Yes | 404
    With pneumococcal vaccination: Yes, Polysaccharide only (PPSV23): number analyzed (Participants) | 404
    With pneumococcal vaccination: Yes, Polysaccharide only (PPSV23) | 180
    With pneumococcal vaccination: Yes, Polysaccharide (PPSV23) + Conjugate (PCV13): number analyzed (Participants) | 404
    With pneumococcal vaccination: Yes, Polysaccharide (PPSV23) + Conjugate (PCV13) | 142
    With pneumococcal vaccination: Yes, Conjugate only (PCV13): number analyzed (Participants) | 404
    With pneumococcal vaccination: Yes, Conjugate only (PCV13) | 82
Conjugate pneumococcal vaccination (PCV13) prior to study inclusion [Count of Participants; unit: Participants] — Overall number of participants, with pneumococcal vaccination, without pneumococcal vaccination is presented. Population: Number Analyzed signifies number of participants evaluable for the specified rows.
  Participants
    Overall: No | 306
    Overall: Yes | 224
    Overall: Yes (Not received influenza vaccine in the same year) | 12
    Overall: Yes (Received influenza vaccine in the same year) | 212
    Without pneumococcal vaccination: No: number analyzed (Participants) | 126
    Without pneumococcal vaccination: No | 126
    Without pneumococcal vaccination: Yes: number analyzed (Participants) | 126
    Without pneumococcal vaccination: Yes | 0
    Without pneumococcal vaccination: Yes (Not received influenza vaccine in the same year): number analyzed (Participants) | 126
    Without pneumococcal vaccination: Yes (Not received influenza vaccine in the same year) | 0
    Without pneumococcal vaccination: Yes (Received influenza vaccine in the same year: number analyzed (Participants) | 126
    Without pneumococcal vaccination: Yes (Received influenza vaccine in the same year | 0
    With pneumococcal vaccination: No: number analyzed (Participants) | 404
    With pneumococcal vaccination: No | 180
    With pneumococcal vaccination: Yes: number analyzed (Participants) | 404
    With pneumococcal vaccination: Yes | 224
    With pneumococcal vaccination: Yes (Not received influenza vaccine in the same year): number analyzed (Participants) | 404
    With pneumococcal vaccination: Yes (Not received influenza vaccine in the same year) | 12
    With pneumococcal vaccination: Yes (Received influenza vaccine in the same year: number analyzed (Participants) | 404
    With pneumococcal vaccination: Yes (Received influenza vaccine in the same year | 212
History of influenza vaccination [Count of Participants; unit: Participants] — Overall number of participants, with pneumococcal vaccination, without pneumococcal vaccination and PCV13 population is presented. Population: Number Analyzed signifies number of participants evaluable for the specified rows.
  Participants
    Overall: No | 57
    Overall: Yes | 473
    Without Pneumococcal Vaccination: number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: No | 48
    Without Pneumococcal Vaccination: Yes | 78
    With Pneumococcal Vaccination: number analyzed (Participants) | 404
    With Pneumococcal Vaccination: No | 9
    With Pneumococcal Vaccination: Yes | 395
    PCV13 Population: number analyzed (Participants) | 114
    PCV13 Population: No | 19
    PCV13 Population: Yes | 95
Most frequent treatments for COPD at baseline [Count of Participants; unit: Participants] — The participants were classified as Yes/No according to pharmacological treatment received for COPD. In the table below, the following have been abbreviated as: Long-Acting Muscarinic Antagonist(LAMA), Long-Acting Beta Agonist(LABA), Inhaled corticosteroid (IC), Short-acting Beta Agonist(SABA), Short Acting Muscarinic Antagonist(SAMA); Phosphodiesterase 4 (PDE4) and N-acetylcysteine(NAC). Overall number of participants, with pneumococcal vaccination, without pneumococcal vaccination and PCV13 population is presented. Population: Number Analyzed signifies number of participants evaluable for the specified rows.
  Participants
    Overall: No | 3
    Overall: Yes | 527
    Overall: Yes (LABA + LAMA) | 237
    Overall: Yes (LAMA) | 143
    Overall: Yes (LABA) | 10
    Overall: Yes (IC + LABA + LAMA) | 173
    Overall: Yes (IC + LABA) | 137
    Overall: Yes (IC + LAMA) | 2
    Overall: Yes (IC+ Theophylline) | 1
    Overall: Yes (SABA) | 221
    Overall: Yes (SAMA) | 35
    Overall: Yes (Others) | 57
    Overall: Yes (PDE4 inhibitors-NAC) | 13
    Overall: Yes (PDE4 inhibitors + LABA + LAMA | 12
    Overall: Yes (PDE4 inhibitors + LAMA) | 7
    Overall: Yes (PDE4 inhibitors + LABA) | 2
    Overall: Yes (Antibiotics-macrolides) | 18
    Overall: Yes (Theophylline + LABA + LAMA) | 5
    Without Pneumococcal Vaccination: No: number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: No | 2
    Without Pneumococcal Vaccination: Yes: number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Yes | 124
    Without Pneumococcal Vaccination: Yes (LABA + LAMA): number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Yes (LABA + LAMA) | 63
    Without Pneumococcal Vaccination: Yes (LAMA): number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Yes (LAMA) | 46
    Without Pneumococcal Vaccination: Yes (LABA): number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Yes (LABA) | 2
    Without Pneumococcal Vaccination: Yes (IC + LABA + LAMA): number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Yes (IC + LABA + LAMA) | 30
    Without Pneumococcal Vaccination: Yes (IC + LABA): number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Yes (IC + LABA) | 42
    Without Pneumococcal Vaccination: Yes (IC + LAMA): number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Yes (IC + LAMA) | 1
    Without Pneumococcal Vaccination: Yes (IC + Theophylline): number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Yes (IC + Theophylline) | 1
    Without Pneumococcal Vaccination: Yes (SABA): number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Yes (SABA) | 58
    Without Pneumococcal Vaccination: Yes (SAMA): number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Yes (SAMA) | 15
    Without Pneumococcal Vaccination: Yes (Others): number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Yes (Others) | 21
    Without Pneumococcal Vaccination: Yes (PDE4 inhibitors-NAC): number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Yes (PDE4 inhibitors-NAC) | 0
    Without Pneumococcal Vaccination: Yes (PDE4 inhibitors + LABA + LAMA): number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Yes (PDE4 inhibitors + LABA + LAMA) | 0
    Without Pneumococcal Vaccination: Yes (PDE4 inhibitors + LAMA): number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Yes (PDE4 inhibitors + LAMA) | 1
    Without Pneumococcal Vaccination: Yes (PDE4 inhibitors + LABA): number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Yes (PDE4 inhibitors + LABA) | 0
    Without Pneumococcal Vaccination: Yes (Antibiotics-Macrolides): number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Yes (Antibiotics-Macrolides) | 3
    Without Pneumococcal Vaccination: Yes (Theophylline + LABA + LAMA): number analyzed (Participants) | 126
    Without Pneumococcal Vaccination: Yes (Theophylline + LABA + LAMA) | 0
    With Pneumococcal Vaccination: No: number analyzed (Participants) | 404
    With Pneumococcal Vaccination: No | 1
    With Pneumococcal Vaccination: Yes: number analyzed (Participants) | 404
    With Pneumococcal Vaccination: Yes | 403
    With Pneumococcal Vaccination: Yes (LABA + LAMA): number analyzed (Participants) | 404
    With Pneumococcal Vaccination: Yes (LABA + LAMA) | 174
    With Pneumococcal Vaccination: Yes (LAMA): number analyzed (Participants) | 404
    With Pneumococcal Vaccination: Yes (LAMA) | 97
    With Pneumococcal Vaccination: Yes (LABA): number analyzed (Participants) | 404
    With Pneumococcal Vaccination: Yes (LABA) | 8
    With Pneumococcal Vaccination: Yes (IC + LABA + LAMA): number analyzed (Participants) | 404
    With Pneumococcal Vaccination: Yes (IC + LABA + LAMA) | 143
    With Pneumococcal Vaccination: Yes (IC + LABA): number analyzed (Participants) | 404
    With Pneumococcal Vaccination: Yes (IC + LABA) | 95
    With Pneumococcal Vaccination: Yes (IC + LAMA): number analyzed (Participants) | 404
    With Pneumococcal Vaccination: Yes (IC + LAMA) | 1
    With Pneumococcal Vaccination: Yes (IC + Theophylline): number analyzed (Participants) | 404
    With Pneumococcal Vaccination: Yes (IC + Theophylline) | 0
    With Pneumococcal Vaccination: Yes (SABA): number analyzed (Participants) | 404
    With Pneumococcal Vaccination: Yes (SABA) | 163
    With Pneumococcal Vaccination: Yes (SAMA): number analyzed (Participants) | 404
    With Pneumococcal Vaccination: Yes (SAMA) | 20
    With Pneumococcal Vaccination: Yes (Others): number analyzed (Participants) | 404
    With Pneumococcal Vaccination: Yes (Others) | 36
    With Pneumococcal Vaccination: Yes (PDE4 inhibitors-NAC): number analyzed (Participants) | 404
    With Pneumococcal Vaccination: Yes (PDE4 inhibitors-NAC) | 13
    With Pneumococcal Vaccination: Yes (PDE4 inhibitors + LABA + LAMA): number analyzed (Participants) | 404
    With Pneumococcal Vaccination: Yes (PDE4 inhibitors + LABA + LAMA) | 12
    With Pneumococcal Vaccination: Yes (PDE4 inhibitors + LAMA): number analyzed (Participants) | 404
    With Pneumococcal Vaccination: Yes (PDE4 inhibitors + LAMA) | 6
    With Pneumococcal Vaccination: Yes (PDE4 inhibitors + LABA): number analyzed (Participants) | 404
    With Pneumococcal Vaccination: Yes (PDE4 inhibitors + LABA) | 2
    With Pneumococcal Vaccination: Yes (Antibiotics-Macrolides): number analyzed (Participants) | 404
    With Pneumococcal Vaccination: Yes (Antibiotics-Macrolides) | 15
    With Pneumococcal Vaccination: Yes (Theophylline + LABA + LAMA): number analyzed (Participants) | 404
    With Pneumococcal Vaccination: Yes (Theophylline + LABA + LAMA) | 5
    PCV13 Population: Yes: number analyzed (Participants) | 114
    PCV13 Population: Yes | 114
    PCV13 Population: Yes (LABA + LAMA): number analyzed (Participants) | 114
    PCV13 Population: Yes (LABA + LAMA) | 52
    PCV13 Population: Yes (LAMA): number analyzed (Participants) | 114
    PCV13 Population: Yes (LAMA) | 39
    PCV13 Population: Yes (LABA): number analyzed (Participants) | 114
    PCV13 Population: Yes (LABA) | 2
    PCV13 Population: Yes (IC + LABA + LAMA): number analyzed (Participants) | 114
    PCV13 Population: Yes (IC + LABA + LAMA) | 34
    PCV13 Population: Yes (Inhaled corticosteroids - IC+ LABA): number analyzed (Participants) | 114
    PCV13 Population: Yes (Inhaled corticosteroids - IC+ LABA) | 29
    PCV13 Population: Yes (IC+ LAMA): number analyzed (Participants) | 114
    PCV13 Population: Yes (IC+ LAMA) | 1
    PCV13 Population: Yes (SABA): number analyzed (Participants) | 114
    PCV13 Population: Yes (SABA) | 49
    PCV13 Population: Yes (SAMA): number analyzed (Participants) | 114
    PCV13 Population: Yes (SAMA) | 8
    PCV13 Population: Yes (Others): number analyzed (Participants) | 114
    PCV13 Population: Yes (Others) | 9
    PCV13 Population: Yes (PDE4 inhibitors: NAC): number analyzed (Participants) | 114
    PCV13 Population: Yes (PDE4 inhibitors: NAC) | 2
    PCV13 Population: Yes (PDE4 inhibitors + LABA + LAMA): number analyzed (Participants) | 114
    PCV13 Population: Yes (PDE4 inhibitors + LABA + LAMA) | 1
    PCV13 Population: Yes (Antibiotics-macrolides): number analyzed (Participants) | 114
    PCV13 Population: Yes (Antibiotics-macrolides) | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Adjusted Rate of Moderate/Severe COPD Exacerbations at Month 24 in PCV 13 Population
Description: COPD exacerbations were defined as a complex of two or more respiratory symptoms (worsening dyspnea, cough, sputum production, chest tightness, or wheezing) related to the underlying COPD, with duration of 3 days or more, that required a change in treatment. Moderate exacerbations were those that required antibiotics and/or systemic corticosteroids without hospitalization. Severe exacerbations were those that lead to hospitalization. Adjusted rate of exacerbation was calculated as (Total number of moderate or severe exacerbations) divided by participant follow-up time in months*24 months.
Time Frame: Baseline and Month 24
Population: PCV13 population included evaluable participants who were administered PCV13 at least 1 month prior providing informed consent to participate in the study and who did not subsequently received PPSV23. All participants reported under "Overall Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row.
Measure: Mean (Standard Deviation); unit: Exacerbation per participant in 24 month
Arm/Group | Participants With COPD
Number analyzed (Participants) | 114
Exacerbation per participant in 24 month | -1.1 (2.5)

2. Primary Outcome: Change in Adjusted Rate of Moderate/Severe Exacerbations by COPD Severity at Month 24 in PCV13 Population
Description: Moderate exacerbations were those that required antibiotics and/or systemic corticosteroids without hospitalization. Severe exacerbations were those that lead to hospitalization. COPD severity was graded as per GOLD criteria. Grade 1 mild/unknown: (FEV1 >= 80 %, FEV1/ FVC < 0.7 or no spirometry data). Grade 2: Moderate: (50% <= FEV1< 80%, FEV1/FVC < 0.7), Grade 3: Severe (30% <=FEV1 < 50%, FEV1/FVC < 0.7), Grade 4: Very severe (FEV1< 30% or FEV1< 50% plus respiratory failure, FEV1/FVC < 0.7). Adjusted rate of exacerbation was calculated as (total no. of moderate or severe exacerbations) divided by participant follow-up time in months*24 months. Change in adjusted rate of moderate/severe exacerbations by COPD severity (Grade 1 and Grade >1) at Month 24 is reported.
Time Frame: Baseline and Month 24
Population: PCV13 population included evaluable participants who were administered PCV13 at least 1 month prior providing informed consent to participate in the study and who did not subsequently received PPSV23. All participants reported under "Overall Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. "Number Analyzed" refers to the number of participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: Exacerbation per participant in 24 month
Arm/Group | Participants With COPD
Number analyzed (Participants) | 114
Exacerbation per participant in 24 month
  Grade 1: Mild/unknown: number analyzed (Participants) | 12
  Grade 1: Mild/unknown | -1.5 (0.9)
  Grade >1: Moderate to Very Severe: number analyzed (Participants) | 102
  Grade >1: Moderate to Very Severe | -1.1 (2.6)

3. Secondary Outcome: Change in Rate of Moderate/Severe COPD Exacerbations at Month 24 in PCV13 Population by History of Influenza Vaccination
Description: Evaluate the impact of influenza and PCV13 vaccination on the reduction of COPD exacerbations. Adjusted rate of exacerbation was calculated as (total number of moderate or severe exacerbations) divided by participant follow-up time in months*24 months. Change in rate of moderate/severe exacerbations with and without history of influenza vaccination is presented in this outcome measure.
Time Frame: Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Exacerbation per participant in 24 month
Arm/Group | Participants With COPD
Number analyzed (Participants) | 114
Exacerbation per participant in 24 month
  Influenza vaccination: No: number analyzed (Participants) | 19
  Influenza vaccination: No | -0.7 (2.2)
  Influenza vaccination: Yes: number analyzed (Participants) | 95
  Influenza vaccination: Yes | -1.2 (2.6)

4. Secondary Outcome: Change From Baseline in Saint George Respiratory Questionnaire (SGRQ) Score at Month 12 and 24 in PCV13 Population
Description: To evaluate the impact of vaccination with PCV13 on patients quality of life SGRQ form was used. It is a self-administered questionnaire developed to measure health status (quality of life) in participants with chronic airflow limitation. The SGRQ consisted of 50 items, where 10 of them were multiple choice and 40 were true or false. Scores were calculated for three domains: Symptoms (eight items; including cough, sputum production, dyspnea or shortness of breath or breathlessness and wheezing, as well as duration, frequency and severity); Activity (16 true or false questions; refers to activities that are limited due to dyspnea);Impacts (26 items; referred to other situations or aspects related to social or psychological functioning affected by the respiratory problems that may alter the participants lifestyle). The total score and scores for each domain ranged from 0 (minimum, best possible health status) to 100 (maximum, worst possible health status).
Time Frame: Baseline, Month 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Participants With COPD
Number analyzed (Participants) | 112
Units on a scale
  Baseline: QOL: number analyzed (Participants) | 108
  Baseline: QOL | 45.7 (15.4)
  Change at Month 12: QOL: number analyzed (Participants) | 82
  Change at Month 12: QOL | -5.6 (17.4)
  Change at Month 24: QOL: number analyzed (Participants) | 77
  Change at Month 24: QOL | -6.0 (13.8)
  Baseline: Symptoms: number analyzed (Participants) | 110
  Baseline: Symptoms | 47.4 (18.9)
  Change at Month 12: Symptoms: number analyzed (Participants) | 87
  Change at Month 12: Symptoms | -9.0 (26.2)
  Change at Month 24: Symptoms: number analyzed (Participants) | 85
  Change at Month 24: Symptoms | -16.3 (23.4)
  Baseline: Activity | 56.3 (21.2)
  Change at Month 12: Activity: number analyzed (Participants) | 85
  Change at Month 12: Activity | -4.6 (19.9)
  Change at Month 24: Activity: number analyzed (Participants) | 79
  Change at Month 24: Activity | -4.2 (17.3)
  Baseline: Impacts | 39.7 (15.4)
  Change at Month 12: Impacts: number analyzed (Participants) | 87
  Change at Month 12: Impacts | -5.6 (19.1)
  Change at Month 24: Impacts: number analyzed (Participants) | 83
  Change at Month 24: Impacts | -6.5 (15.5)

5. Secondary Outcome: Change From Baseline in COPD Assessment Test (CAT) Score at Month 12 and 24 in PCV13 Population
Description: To evaluate the impact of vaccination with PCV13 on patients quality of life ,CAT questionnaire is used. It is used to measure the impact COPD on the participant's wellbeing and daily life and severity of symptoms. The CAT has 8 questions, with score ranging from 0 to 5 for each question, where 0 = no impairment and 5=severe impairment. Total score was calculated as the sum of scores of individual questions and ranged from 0 to 40 with higher scores indicating more severe disease.
Time Frame: Baseline, Month 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Participants With COPD
Number analyzed (Participants) | 109
Units on a scale
  Baseline | 15.5 (7.5)
  Change at Month 12: number analyzed (Participants) | 85
  Change at Month 12 | -1.7 (6.3)
  Change at Month 24: number analyzed (Participants) | 80
  Change at Month 24 | -1.8 (6.1)

6. Secondary Outcome: Change From Baseline in Forced Expiratory Volume (FEV1) at Month 24 in PCV13 Population
Description: To evaluate the impact of vaccination with PCV13 on the decrease of FEV1 was evaluated. FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration.
Time Frame: Baseline, Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Participants With COPD
Number analyzed (Participants) | 114
Percentage
  Baseline | 51.9 (19.0)
  Change at Month 24 | -1.7 (10.9)

7. Secondary Outcome: Percentage of Participants With COPD Vaccinated With PCV13
Description: Percentage of evaluable study participants vaccinated with PCV13 prior or after inclusion in the study.
Time Frame: Up to Month 24
Population: Evaluable Population according to inclusion criteria (at least 2 years of clinical history available that includes records of previous moderate/severe exacerbations, influenza and pneumococcal vaccination history comorbidities and previous treatments). The participants were administered PCV13 at least 2 years before or after giving informed consent
Measure: Number; unit: Percentage of Participants
Arm/Group | Participants With COPD
Number analyzed (Participants) | 530
Percentage of Participants | 46.8

8. Other Pre Specified Outcome: Mean Cost Saving Per COPD Participant With PCV13
Description: Overall cost of hospitalization and/or treatment of exacerbation episode based on days of hospitalization or Intensive care unit and treatment received were planned to be analyzed in this outcome measure.
Time Frame: Up to Month 24
Population: PCV13 population included evaluable participants that were administered PCV13 at least 1 month prior providing informed consent to participate in the study and that did not subsequently received PPSV23.
Measure: Number; unit: Euro per participant per year
Arm/Group | Participants With COPD
Number analyzed (Participants) | 114
Euro per participant per year | NA — Cost saving could not be calculated as unitary cost was not reported.

ADVERSE EVENTS:
Time Frame: Up to 24 months
Description: Same event may appear as both an AE and Serious Adverse Events (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Participants With COPD
All-Cause Mortality (participants affected / at risk) | 39/530
Serious Adverse Events (participants affected / at risk) | 78/530
Other Adverse Events (participants affected / at risk) | 10/530
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With COPD (N=530)
Pneumonia (Infections and infestations) | 17
COVID-19 pneumonia (Infections and infestations) | 10
COVID-19 (Infections and infestations) | 3
Abdominal sepsis (Infections and infestations) | 1
Appendicitis perforated (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Klebsiella bacteraemia (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Peritonitis bacterial (Infections and infestations) | 1
Pneumonia staphylococcal (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Cardio-respiratory arrest (Cardiac disorders) | 6
Cardiac failure (Cardiac disorders) | 4
Acute myocardial infarction (Cardiac disorders) | 3
Cardiac failure congestive (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Death (General disorders) | 9
Sudden death (General disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Encephalopathy (Nervous system disorders) | 1
Guillain-Barre syndrome (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Shock (Vascular disorders) | 1
Bicytopenia (Blood and lymphatic system disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Lung operation (Surgical and medical procedures) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With COPD (N=530)
Chest pain (General disorders) | 1
Local reaction (General disorders) | 1
Vaccination site reaction (General disorders) | 1
COVID-19 (Infections and infestations) | 1
COVID-19 pneumonia (Infections and infestations) | 1
Tachyarrhythmia (Cardiac disorders) | 1
Immunosuppression (Immune system disorders) | 1
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary resection (Surgical and medical procedures) | 1

LIMITATIONS AND CAVEATS:
Several limitations related to the study, such as lack of data about relevant confounding factors, and a lower than expected sample size, which makes impossible the adjustment of analyses by relevant confounding factors such as age, presence and number of comorbidities, severity of the disease, etc, make difficult to discard that the changes in the exacerbation rates are due to other causes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-10-31): https://cdn.clinicaltrials.gov/large-docs/54/NCT03276754/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/54/NCT03276754/SAP_001.pdf